CLINICAL TRIAL: NCT05558527
Title: Effects of Trauma and Discrimination on the Social Regulation of Threat-related Vigilance and Arousal
Brief Title: The Social Regulation of Threat-related Vigilance and Arousal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1883993-2
Record Dates: First submitted 2022-08-12; First posted 2022-09-28 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Psychological Trauma, Historical; Discrimination, Racial; Emotion Regulation; Social Interaction; Hypervigilance; Anxiety
Keywords: psychological trauma; ethnoracial discrimination; hypervigilance; anticipated threat; social emotion regulation; social touch
MeSH Terms: conditions — Historical Trauma; Racism; Emotional Regulation; Anxiety Disorders; Psychological Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social support from a romantic partner (Experimental): Participants will hold the hand of their romantic partner
  Interventions: Behavioral: social support
- Social support from a stranger (Active Comparator): Participants will hold the hand of a stranger
  Interventions: Behavioral: social support
- No social support (No Intervention): Participants will hold a stress ball

INTERVENTIONS:
Behavioral: social support — social support is provided in the form of social touch (hand holding)
  Arms: Social support from a romantic partner; Social support from a stranger

SUMMARY:
This study will examine the effects of social support on threat vigilance and arousal using eye tracking. We will also test the moderating effects of trauma and discrimination history.

DETAILED DESCRIPTION:
Both interpersonal trauma (IPT) and ethno-racial discrimination amplify risk for hyper-arousal symptoms of posttraumatic stress disorder (PTSD), but the mechanism of this effect is unclear. Prior research suggests that social support plays an important role in regulating emotional responses, a process called social emotion regulation. This study will test whether a history of IPT and/or ethno-racial discrimination influence the social regulation of arousal and vigilance. Social regulation will be tested by contrasting responses under conditions with and without social support.

ELIGIBILITY:
Inclusion Criteria:

* In a stable romantic relationship for 6 months or more
* Normal vision or corrected-to-normal vision
* Fluent in English

Exclusion Criteria:

* If vision is corrected-to-normal, needs to use hard contact lenses, bifocal contact lenses, or glasses
* Experienced a traumatic event within the past 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Vigilance Related Eye Movements - Number of Eye Fixations | Collected from minute 15 to minute 45 of study participation, approximately
  Participants will view 15 pictures of natural environmental scenes for 10 seconds per image. We will use an eye tracker to examine the number of eye fixations per scene. A greater number of fixations during the 10 second presentation of a scene would indicate greater vigilance.
Vigilance Related Eye Movements - Visual Scanning | Collected from minute 15 to minute 45 of study participation, approximately
  Participants will view 15 pictures of natural environmental scenes for 10 seconds per image. We will use an eye tracker to examine the proportion of the scene that they look at (fixate on) out of approximately 80 possible sectors. A greater proportion of the scene they fixate on would indicate greater vigilance.
Threat-Related Physiological Arousal - Pupil Dilation | Collected from minute 45 to minute 75 of study participation, approximately
  Participants will view a series of visual cues (either an 'X' or an 'O') where an 'X' signals a possible (20% probability) aversive auditory stimulus (human scream). We will examine pupil dilation during the task in order to measure arousal in response to uncertain threat. We will calculate average pupil dilation during the wait period after threat cues (X) and after safety cues (O). We will subtract average pupil dilation after safety cues from threat cues to create an index of threat-related arousal. Greater pupil dilation (for threat minus safety cues) would indicate greater threat-related arousal.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L Lancaster, PhD, Principal Investigator — University of Nevada, Reno
Locations (1):
- University of Nevada, Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data including primary and secondary outcomes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: within 6 months after publication
Access Criteria: email request to the study PI (cynthialancaster@unr.edu)